CLINICAL TRIAL: NCT00461110
Title: A Phase 1 Study of BMS-663513 in Combination With Chemoradiation in Subjects With Non Small Cell Lung Carcinoma (NSCLC)
Brief Title: A Study of BMS-663513 in Combination With Chemoradiation in Subjects With Non Small Cell Lung Carcinoma (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA186-005
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — urelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Active
  Interventions: Drug: BMS-663513
- 2 (Experimental): Active
  Interventions: Drug: BMS-663513

INTERVENTIONS:
Drug: BMS-663513 — mg/kg, IV, 0.3, 1,3,6,10 mg/kg, q 3 wks, 12 weeks
  Other Names: Anti-CD137

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and assess the safety and tolerability of escalating doses of BMS-663513 when given in combination with either radiotherapy alone or radiotherapy plus paclitaxel and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC who are eligible to receive a 6 week course of RT
* Part 1 - not candidates for definitive RT
* Part 2 - candidates for definitive RT

Exclusion Criteria:

* Severe COPD, pulmonary infection or interstitial pneumonitis
* Recent cellulitis
* Autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
To determine the MTD and assess safety and tolerability of single ascending doses of BMS-663513 when given in combination with radiotherapy alone or radiotherapy plus paclitaxel and carboplatin to subjects with Non Small Cell Lung Carcinoma | throughout the study

SECONDARY OUTCOMES:
Assess the PKs of BMS-663513 and the effect of BMS-663513 on immune system markers | end of study
Describe anti-tumor activity | throughout the study
Obtain blood and plasma for exploratory research | several timepoints throughout the study
Obtain archival tissue for predictive marker research | at screening

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - The Cancer Institute Of New Jersey, New Brunswick, New Jersey
  - Nyu Clinical Cancer Center, New York, New York
  - Thomas Jefferson Univ Hospital, Philadelphia, Pennsylvania
  - University Of Texas Southwestern Medical Center, Dallas, Texas